CLINICAL TRIAL: NCT07402772
Title: Performance of the Osteoporosis Self-Assessment Tool (OST) and Osteoporosis Risk Assessment Index (ORAI) in Predicting Osteoporosis in Postmenopausal Turkish Women
Brief Title: Female Osteoporosis
Acronym: OST and ORAI
Status: Not yet recruiting | Type: Observational
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Fatma Gül Ülkü Demir, MD, Kayseri City Hospital
Other Study IDs: Female osteoporosis
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-10

CONDITIONS: Female Osteoporosis
Keywords: female osteoporosis; OST; ORAI

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- female osteoporosis group

SUMMARY:
The aim of this study is to compare the Osteoporosis Risk Assessment Tool and the Osteoporosis Self-Assessment Tool with the gold standard DEXA in determining the risk of osteoporosis in the lumbar and femoral regions in female individuals in the Turkish population, and to investigate their sensitivity and specificity in the first stage of screening for the detection of female osteoporosis.

DETAILED DESCRIPTION:
This study will be conducted as a single-center, retrospective study at the Physical Medicine and Rehabilitation Clinic of Kayseri City Hospital between January 2024 and January 2025. This study will include female patients aged 50-75 who underwent osteoporosis screening with DEXA at the Kayseri City Hospital FTR outpatient clinics between January 2021 and January 2024. Patient data will be obtained retrospectively from the hospital database. Sociodemographic data (age, height, weight, body mass index) and current laboratory data (complete blood count, biochemical values (fasting blood sugar, BUN, creatinine, AST, ALT, calcium, phosphorus, alkaline phosphatase, total protein, albumin, parathyroid hormone, vitamin D3, T4, TSH), and DEXA values (bone mineral density, lumbar vertebrae, and femoral neck and total femur T scores) will be recorded. The OST score will be calculated using body weight and age parameters. The ORAI score will be calculated using age, weight, and estrogen use from hospital data.

The data will be evaluated using the SPSS 24.0 software package. Descriptive statistical analyses will include calculations of mean, standard deviation, frequency, and percentages. In comparative statistics, the Student T-test or Mann Whitney U-test will be used to compare independent groups. Chi-square analysis will be applied to compare categorical variables. Pearson or Spearman correlation analyses will be applied to evaluate the relationship between variables. Both groups will be compared, and p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion criteria:

* Postmenopausal women aged 50-75
* Patients who underwent imaging with the STRATOS DEXA device at Kayseri City Hospital

Exclusion criteria:

* Patients younger than 50 or older than 75 years of age
* Patients with secondary osteoporosis
* Male patients
* Patients with uncontrolled severe comorbid conditions
* Patients with a history of pathological fractures

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender female participant
Study Population: This study will include female patients aged 50-75 who underwent osteoporosis screening with DEXA at the Kayseri City Hospital FTR outpatient clinics between January 2021 and January 2024.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2026-02-04 (Estimated); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Dual-energy X-ray absorptiometry (DEXA) | January 2021 - January 2024
  Dual-energy X-ray absorptiometry (DEXA)
Osteoporosis Self-Assessment Tool (OST) | January 2021 - January 2024
  Osteoporosis Self-Assessment Tool (OST)
Osteoporosis Risk Assessment Index (ORAI) | January 2021 - January 2024
  Osteoporosis Risk Assessment Index (ORAI)

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Gül ÜLKÜ DEMİR, MD, Principal Investigator — Kayseri City Hospital

IPD SHARING:
Plan to Share IPD: Undecided
There is not a plan to make IPD available.